CLINICAL TRIAL: NCT01624207
Title: A Multi-center, Randomized, Open-labeled Clinical Trial to Evaluate Efficacy and Safety of Atorva® 20mg Versus Lipitor® 20mg in Korean Patients With Hypercholesterolemia
Brief Title: The Efficacy and Safety of Atorva® 20mg Versus Lipitor® 20mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Yuhan corp., Seoul, Korea (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROYAL; H-1002-038-309 (Other: Seoul National University Hospital)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Hypercholesterolemia
Keywords: Atorva; generic; atorvastatin; hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorva (Experimental): generic formulation (Atorva®) of atorvastatin 20mg once daily
  Interventions: Drug: generic formulation of atorvastatin (Atorva®)
- Lipitor (Active Comparator): branded formulation (Lipitor®) of atorvastatin 20mg once daily
  Interventions: Drug: branded formulation of atorvastatin (Lipitor®)

INTERVENTIONS:
Drug: generic formulation of atorvastatin (Atorva®) — Treatment with generic formulation of atorvastatin (Atorva®) once daily, for 8 weeks
  Arms: Atorva
Drug: branded formulation of atorvastatin (Lipitor®) — Treatment with branded formulation of atorvastatin (Lipitor®)once daily, for 8 weeks
  Arms: Lipitor

SUMMARY:
The generic formulation of atorvastatin (Atorva®) 20mg was not inferior to the branded formulation of atorvastatin (Lipitor®) 20mg in this 8-week treatment of hyperlipidemic Korean patients. In PP analysis, the LDL cholesterol goal achievement rate was significantly higher in Atorva group. Both treatments were well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were men or women aged between 20 and 79 years who have not achieved LDL cholesterol goals using the National Cholesterol Education Program Adult Treatment Panel Ⅲ (NCEP-ATP Ⅲ) guideline, with the treatment goal of LDL cholesterol being <100 mg/dL for patients with coronary artery disease (CAD) or CAD-equivalent disease, <130 mg/dL for patients with multiple risk factors (10-year coronary heart disease [CHD] risk ≤20%), and <160 mg/dL for patients with 0 to 1 risk factors.

Exclusion Criteria:

* Exclusion criteria were as follows: currently taking any kind of anti-hyperlipidemic drug (within 4 weeks before enrollment); hypersensitivity or intolerance to atorvastatin or other HMG-CoA reductase inhibitor; newly diagnosed (within 3 months before enrollment) or uncontrolled diabetes (hemoglobin A1C >9%); uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg); hepatic dysfunction (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] levels ≥2 times the upper limit of normal [ULN]); an unexplained serum creatinine kinase (CK) elevation >2 times the ULN, chronic renal failure (a serum creatinine concentration >2.5 mg/dL); in patients who experienced operation at the time of screening, the patients must have a result of lipid profiles within 24 hours or after 6 weeks; a history of malignancy or cervical dysplasia; pregnant or breastfeeding women; women of childbearing potential had to be using adequate methods of contraception; a history of drug abuse or alcoholism; participation in other studies 4 weeks before enrollment. Patients could also be excluded if their participation was considered inappropriate by the study physician.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
% change of LDL cholesterol | After 8 weeks of treatment
  The difference in percent change of serum LDL cholesterol concentration between genericAtorva and Lipitor branded group

SECONDARY OUTCOMES:
% change of other lipid paramenters(total cholesterol, high-density lipoprotein [HDL] cholesterol, triglyceride [TG], apolipoprotein B [ApoB] and apolipoprotein A1 [ApoA1]) | After 8 weeks of treatment
% change of lipoprotein and apolipoprotein ratios (ApoB/ApoA1 ratio, total cholesterol/HDL cholesterol ratio) | After 8 weeks of treatment
Change of highly sensitive C-reactive protein (hsCRP) | After 8 weeks of treatment
LDL cholesterol goal achievement rate | After 8 weeks of treatment
  LDL cholesterol goal achievement rate according to NECP-ATP III guideline

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea